CLINICAL TRIAL: NCT02242045
Title: A Phase 1b Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Idelalisib in Japanese Subjects With Relapsed or Refractory Indolent B-Cell Non-Hodgkin Lymphomas or Chronic Lymphocytic Leukemia
Brief Title: Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Idelalisib in Japanese Participants With Relapsed or Refractory Indolent B-Cell Non-Hodgkin Lymphomas (iNHL) or Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-313-1380
Expanded Access: NCT02136511 (Approved for marketing)
Record Dates: First submitted 2014-09-13; First posted 2014-09-16 (Estimated); Results first posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-02

CONDITIONS: Chronic Lymphocytic Leukemia; Indolent Non-Hodgkin Lymphoma; Follicular Lymphoma; Small Lymphocytic Lymphoma; Lymphoplasmacytic Lymphoma (With or Without Waldenstrom Macroglobulinemia); Marginal Zone Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — idelalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Idelalisib (Experimental): Participants with iNHL or CLL will receive idelalisib until the earliest of the following: unacceptable toxicity, substantial noncompliance, disease progression, pregnancy, initiation of another anticancer or experimental therapy, investigator discretion, or idelalisib discontinuation.
  Interventions: Drug: Idelalisib

INTERVENTIONS:
Drug: Idelalisib — 150 mg tablet(s) administered orally twice daily
  Other Names: Zydelig®; GS-1101; CAL-101

SUMMARY:
The primary objective of this study is to evaluate the 28-day safety and tolerability, and to determine the pharmacokinetics (PK) of idelalisib in Japanese participants with relapsed or refractory indolent B-cell non-Hodgkin lymphomas (iNHL) or chronic lymphocytic leukemia (CLL).

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with mature B-cell malignancies of iNHL including follicular lymphoma, small lymphocytic lymphoma, lymphoplasmacytic lymphoma, marginal zone lymphoma, and CLL by World Health Organization classification
* Must have been born in Japan and must not have lived outside of Japan for > 1 year in the 5 years prior to Day 1
* Must be able to trace maternal and paternal ancestry of parents and grandparents as Japanese
* Must have been previously treated with at least 1 regimen for iNHL or CLL and currently require treatment
* Discontinuation of all therapy (including radiotherapy, chemotherapy, immunotherapy, or investigational therapy) for the treatment of iNHL or CLL ≥ 4 weeks prior to Day 1
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Required baseline laboratory data (within 4 weeks prior to Day 1)
* A negative serum pregnancy test for female participants of childbearing potential
* Males and females of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception.
* In the judgment of the investigator, participation in the protocol offers an acceptable benefit-to-risk ratio when considering current disease status, medical condition, and the potential benefits and risks of alternative treatments for the individual's disease.

Key Exclusion Criteria:

* Known histological transformation to an aggressive histology
* Known presence of myelodysplastic syndrome
* History of iNHL or CLL with central nervous system involvement
* Life expectancy < 120 days as per investigator assessment
* History of a nonlymphoid malignancy with the following exceptions:

  * the malignancy has been in remission without treatment for ≥ 5 years prior to Day 1, or
  * carcinoma in situ of the cervix, or
  * adequately treated basal or squamous cell skin cancer or other localized nonmelanoma skin cancer, or
  * surgically treated low-grade prostate cancer, or
  * ductal carcinoma in situ of the breast treated with lumpectomy alone
* On-going drug-induced liver injury, alcoholic liver disease, nonalcoholic steatohepatitis, primary biliary cirrhosis, extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver, or portal hypertension
* History or diagnosis of pneumonitis or interstitial lung disease.
* On-going inflammatory bowel disease
* Pregnancy or breastfeeding
* History of prior allogeneic hematopoietic stem cell or solid organ transplantation
* Concurrent participation in another therapeutic clinical trial
* Prior or on-going clinically significant illness, medical condition, surgical history, physical finding, electrocardiogram finding, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the individual or impair the assessment of study results.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2014-12-25 (Actual); Study Completion 2017-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (3):
- Japan (3):
  - Aichi
  - Miyagi
  - Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Kinoshita T, Fukuhara N, Nagai H, Izutsu K, Kobayashi Y, et al. Phase 1b and Pharmacokinetic Study of Idelalisib in Japanese Patients with Relapsed or Refractory (R/R) Indolent B-Cell Non-Hodgkin Lymphoma (iNHL) or Chronic Lymphocytic Leukemia (CLL) [Abstract 85914]. Blood 2015;126:5089
- [Result] Fukuhara N, Kinoshita T, Yamamoto K, Nagai H, Izutsu K, Yamamoto G, Bhargava P, Rajakumaraswamy N, Humeniuk R, Mathias A, Xing G, Fukui M, Tobinai K. Phase 1b study to investigate the safety and tolerability of idelalisib in Japanese patients with relapsed/refractory follicular lymphoma and chronic lymphocytic leukemia. Jpn J Clin Oncol. 2020 Dec 16;50(12):1395-1402. doi: 10.1093/jjco/hyaa153. PMID 32856068

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Japan. The first participant was screened on 01 October 2014. The last study visit occurred on 17 October 2017.
Pre-assignment Details: 6 participants were screened.
Groups:
- Idelalisib: Participants with indolent non-hodgkin lymphoma (iNHL) or chronic lymphocytic leukemia (CLL) received idelalisib 150 mg tablet orally twice daily until the earliest of the following: unacceptable toxicity, substantial noncompliance, disease progression, pregnancy, initiation of another anticancer or experimental therapy, investigator discretion, or idelalisib discontinuation.
Period: Overall Study
Arm/Group | Idelalisib
Started | 6
Completed | 0
Not Completed | 6
Not completed — Investigator's Discretion | 1
Not completed — Progressive Disease | 2
Not completed — Unable to tolerate rechallenge with idelalisib | 1
Not completed — Initiated another anti-cancer or experimental therapy | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- Idelalisib: Participants with iNHL or CLL received idelalisib 150 mg tablet orally twice daily until the earliest of the following: unacceptable toxicity, substantial noncompliance, disease progression, pregnancy, initiation of another anticancer or experimental therapy, investigator discretion, or idelalisib discontinuation.
Arm/Group | Idelalisib
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) Within 28 Days of Idelalisib Exposure
Description: An AE was any untoward medical occurrence in a clinical study participant which did not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAEs were defined as 1 or both of the following: 1) Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug; and/or 2) Any AEs leading to premature discontinuation of study drug.
Time Frame: First dose date up to 28 days
Population: The Full Analysis Set included all participants who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Idelalisib
Number analyzed (Participants) | 6
percentage of participants
  TEAEs | 66.7
  SAEs | 16.7

2. Primary Outcome: Percentage of Participants Experiencing TEAEs Related to Idelalisib Within 28 Days of Idelalisib Exposure
Description: as for outcome 1
Time Frame: First dose date up to 28 days
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Idelalisib
Number analyzed (Participants) | 6
percentage of participants | 0

3. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities Within 28 Days of Idelalisib Exposure by Worst Grade at Postbaseline
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least one toxicity grade from baseline. If the relevant baseline laboratory value was missing, then any abnormality of at least Grade 1 observed within the time frame specified above was considered treatment-emergent.The most severe graded abnormality from all tests was counted for each participant. Treatment-emergent laboratory abnormalities were graded per Common Terminology Criteria for Adverse Events (CTCAE), Version 4.03 where 1=Mild, 2=Moderate, 3=Severe, 4=Potentially Life Threatening.
Time Frame: First dose date up to 28 days
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Idelalisib
Number analyzed (Participants) | 6
percentage of participants
  Leukocytosis (Grade 1) | 0
  Leukocytosis (Grade 2) | 0
  Leukocytosis (Grade 3) | 16.7
  Leukocytosis (Grade 4) | 0
  White blood cell decreased (Grade 1) | 16.7
  White blood cell decreased (Grade 2) | 0
  White blood cell decreased (Grade 3) | 16.7
  White blood cell decreased (Grade 4) | 0
  Neutrophil count decreased (Grade 1) | 16.7
  Neutrophil count decreased (Grade 2) | 16.7
  Neutrophil count decreased (Grade 3) | 0
  Neutrophil count decreased (Grade 4) | 0
  Hypocalcemia (Grade 1) | 0
  Hypocalcemia (Grade 2) | 16.7
  Hypocalcemia (Grade 3) | 0
  Hypocalcemia (Grade 4) | 0
  Cholesterol high (Grade 1) | 33.3
  Cholesterol high (Grade 2) | 0
  Cholesterol high (Grade 3) | 0
  Cholesterol high (Grade 4) | 0
  Creatinine increased (Grade 1) | 16.7
  Creatinine increased (Grade 2) | 0
  Creatinine increased (Grade 3) | 0
  Creatinine increased (Grade 4) | 0
  Chronic Kidney Disease (Grade 1) | 0
  Chronic Kidney Disease (Grade 2) | 33.3
  Chronic Kidney Disease (Grade 3) | 0
  Chronic Kidney Disease (Grade 4) | 0
  Hypertriglyceridemia (Grade 1) | 33.3
  Hypertriglyceridemia (Grade 2) | 16.7
  Hypertriglyceridemia (Grade 3) | 0
  Hypertriglyceridemia (Grade 4) | 0

4. Primary Outcome: Percentage of Participants Who Permanently Discontinued Idelalisib Due to a TEAE Within 28 Days of Idelalisib Exposure
Description: as for outcome 1
Time Frame: First dose date up to 28 days
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Idelalisib
Number analyzed (Participants) | 6
percentage of participants | 0

5. Primary Outcome: Plasma Concentration of Idelalisib and Its Major Metabolite GS-563117 on Day 1
Description: Lower limit of quantitation was 5 ng/mL for idelalisib and metabolite GS-563117 both.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose on Day 1
Population: The Pharmacokinetic (PK) Analysis Set included all enrolled participants who took at least 1 dose of study drug and had at least 1 nonmissing postdose value reported by the PK laboratory.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Idelalisib
Number analyzed (Participants) | 6
ng/mL
  Idelalisib: Predose | NA (NA) — Values were all below the limit of quantitation.
  Idelalisib: 0.5 hour | 188.4 (322.97)
  Idelalisib: 1 hour | 763.9 (1141.85)
  Idelalisib: 1.5 hour | 1454.0 (1255.23)
  Idelalisib: 2 hour | 2097.4 (1483.25)
  Idelalisib: 3 hour | 2226.5 (1231.66)
  Idelalisib: 4 hour | 2042.3 (1048.57)
  Idelalisib: 6 hour | 1215.0 (797.50)
  Idelalisib: 8 hour | 718.5 (532.06)
  Idelalisib: 12 hour | 291.4 (247.66)
  GS-563117: Predose | NA (NA) — Values were all below the limit of quantitation.
  GS-563117: 0.5 hour | 6.38 (7.095)
  GS-563117: 1 hour | 134.92 (153.644)
  GS-563117: 1.5 hour | 478.75 (507.114)
  GS-563117: 2 hour | 1005.12 (781.188)
  GS-563117: 3 hour | 2011.00 (1206.687)
  GS-563117: 4 hour | 2121.00 (1352.570)
  GS-563117: 6 hour | 2288.33 (1358.446)
  GS-563117: 8 hour | 2195.00 (1494.054)
  GS-563117: 12 hour | 1677.83 (1307.384)

6. Primary Outcome: Plasma Concentration of Idelalisib and Its Major Metabolite GS-563117 on Day 8
Time Frame: Predose and 1.5 hours postdose on Day 8
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Idelalisib
Number analyzed (Participants) | 6
ng/mL
  Idelalisib: Predose | 463.2 (220.75)
  Idelalisib: 1.5 hour | 2138.5 (759.23)
  GS-563117: Predose | 2703.33 (1866.555)
  GS-563117: 1.5 hour | 3040.00 (1736.237)

7. Primary Outcome: Plasma Concentration of Idelalisib and Its Major Metabolite GS-563117 on Day 15
Time Frame: Predose and 1.5 hours postdose on Day 15
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Idelalisib
Number analyzed (Participants) | 6
ng/mL
  Idelalisib: Predose | 459.3 (203.64)
  Idelalisib: 1.5 hour | 2648.3 (1601.70)
  GS-563117: Predose | 3326.67 (2655.234)
  GS-563117: 1.5 hour | 3636.67 (2547.883)

8. Primary Outcome: Plasma Concentration of Idelalisib and Its Major Metabolite GS-563117 on Day 22
Time Frame: Predose and 1.5 hours postdose on Day 22
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Idelalisib
Number analyzed (Participants) | 6
ng/mL
  Idelalisib: Predose | 358.7 (237.86)
  Idelalisib: 1.5 hour | 2155.0 (782.73)
  GS-563117: Predose | 2318.33 (1070.111)
  GS-563117: 1.5 hour | 2828.33 (1749.153)

9. Primary Outcome: Plasma Concentration of Idelalisib and Its Major Metabolite GS-563117 on Day 29
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose on Day 29
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Idelalisib
Number analyzed (Participants) | 6
ng/mL
  Idelalisib: Predose | 501.2 (329.02)
  Idelalisib: 0.5 hour | 666.8 (454.58)
  Idelalisib: 1 hour | 1107.8 (891.69)
  Idelalisib: 1.5 hour | 1523.3 (990.84)
  Idelalisib: 2 hour | 1940.0 (1028.47)
  Idelalisib: 3 hour | 2313.3 (644.13)
  Idelalisib: 4 hour | 1843.8 (701.36)
  Idelalisib: 6 hour | 1141.2 (509.70)
  Idelalisib: 8 hour | 707.2 (340.26)
  Idelalisib: 12 hour | 403.0 (315.41)
  GS-563117: Predose Day 29 | 3075.00 (2546.698)
  GS-563117: 0.5 hour | 2913.33 (2855.182)
  GS-563117: 1 hour | 2833.33 (2535.387)
  GS-563117: 1.5 hour | 2930.00 (2585.660)
  GS-563117: 2 hour | 3185.00 (2799.691)
  GS-563117: 3 hour | 3781.67 (3058.283)
  GS-563117: 4 hour | 3893.33 (2996.309)
  GS-563117: 6 hour | 3653.33 (2900.232)
  GS-563117: 8 hour | 3428.33 (2987.376)
  GS-563117: 12 hour | 2871.67 (3309.601)

10. Secondary Outcome: Percentage of Participants Experiencing TEAEs and SAEs Beyond 28 Days of Idelalisib Exposure
Description: as for outcome 1
Time Frame: First dose date up to 30 days after last dose (up to approximately 3 years)
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Idelalisib
Number analyzed (Participants) | 6
percentage of participants
  TEAEs | 100.0
  SAEs | 83.3

11. Secondary Outcome: Percentage of Participants Experiencing TEAEs Related to Idelalisib Beyond 28 Days of Idelalisib Exposure
Description: as for outcome 1
Time Frame: First dose date up to 30 days after last dose (up to approximately 3 years)
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Idelalisib
Number analyzed (Participants) | 6
percentage of participants | 83.3

12. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities Beyond 28 Days of Idelalisib Exposure by Worst Grade at Postbaseline
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least one toxicity grade from baseline. The most severe graded abnormality from all tests was counted for each participant. Treatment-emergent laboratory abnormalities were graded per CTCAE, Version 4.03 where 1=Mild, 2=Moderate, 3=Severe, 4=Potentially Life Threatening.
Time Frame: First dose date up to 30 days after last dose (up to approximately 3 years)
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Idelalisib
Number analyzed (Participants) | 6
percentage of participants
  Anemia (Grade 1) | 0
  Anemia (Grade 2) | 16.7
  Anemia (Grade 3) | 0
  Anemia (Grade 4) | 0
  Leukocytosis (Grade 1) | 0
  Leukocytosis (Grade 2) | 0
  Leukocytosis (Grade 3) | 16.7
  Leukocytosis (Grade 4) | 0
  White blood cell decreased (Grade 1) | 50.0
  White blood cell decreased (Grade 2) | 0
  White blood cell decreased (Grade 3) | 16.7
  White blood cell decreased (Grade 4) | 0
  Lymphocyte count decreased (Grade 1) | 0
  Lymphocyte count decreased (Grade 2) | 16.7
  Lymphocyte count decreased (Grade 3) | 16.7
  Lymphocyte count decreased (Grade 4) | 0
  Neutrophil count decreased (Grade 1) | 33.3
  Neutrophil count decreased (Grade 2) | 16.7
  Neutrophil count decreased (Grade 3) | 33.3
  Neutrophil count decreased (Grade 4) | 0
  Alanine aminotransferase increased (Grade 1) | 33.3
  Alanine aminotransferase increased (Grade 2) | 0
  Alanine aminotransferase increased (Grade 3) | 0
  Alanine aminotransferase increased (Grade 4) | 16.7
  Hypoalbuminemia (Grade 1) | 0
  Hypoalbuminemia (Grade 2) | 16.7
  Hypoalbuminemia (Grade 3) | 0
  Hypoalbuminemia (Grade 4) | 0
  Hypocalcemia (Grade 1) | 0
  Hypocalcemia (Grade 2) | 16.7
  Hypocalcemia (Grade 3) | 0
  Hypocalcemia (Grade 4) | 0
  Alkaline phosphatase increased (Grade 1) | 16.7
  Alkaline phosphatase increased (Grade 2) | 0
  Alkaline phosphatase increased (Grade 3) | 0
  Alkaline phosphatase increased (Grade 4) | 0
  Aspartate aminotransferase increased (Grade 1) | 33.3
  Aspartate aminotransferase increased (Grade 2) | 0
  Aspartate aminotransferase increased (Grade 3) | 16.7
  Aspartate aminotransferase increased (Grade 4) | 0
  Blood bilirubin increased (Grade 1) | 16.7
  Blood bilirubin increased (Grade 2) | 0
  Blood bilirubin increased (Grade 3) | 0
  Blood bilirubin increased (Grade 4) | 0
  Cholesterol high (Grade 1) | 16.7
  Cholesterol high (Grade 2) | 16.7
  Cholesterol high (Grade 3) | 0
  Cholesterol high (Grade 4) | 0
  Creatinine increased (Grade 1) | 50.0
  Creatinine increased (Grade 2) | 16.7
  Creatinine increased (Grade 3) | 0
  Creatinine increased (Grade 4) | 0
  Chronic Kidney Disease (Grade 1) | 0
  Chronic Kidney Disease (Grade 2) | 50.0
  Chronic Kidney Disease (Grade 3) | 16.7
  Chronic Kidney Disease (Grade 4) | 0
  Gamma Glutamyl Transferase increased (Grade 1) | 50.0
  Gamma Glutamyl Transferase increased (Grade 2) | 16.7
  Gamma Glutamyl Transferase increased (Grade 3) | 0
  Gamma Glutamyl Transferase increased (Grade 4) | 0
  Hyperglycemia (Grade 1) | 50.0
  Hyperglycemia (Grade 2) | 0
  Hyperglycemia (Grade 3) | 16.7
  Hyperglycemia (Grade 4) | 0
  Hypophosphatemia (Grade 1) | 0
  Hypophosphatemia (Grade 2) | 16.7
  Hypophosphatemia (Grade 3) | 33.3
  Hypophosphatemia (Grade 4) | 0
  Hypokalemia (Grade 1) | 0
  Hypokalemia (Grade 2) | 0
  Hypokalemia (Grade 3) | 16.7
  Hypokalemia (Grade 4) | 16.7
  Hyponatremia (Grade 1) | 33.3
  Hyponatremia (Grade 2) | 0
  Hyponatremia (Grade 3) | 0
  Hyponatremia (Grade 4) | 0
  Hypertriglyceridemia (Grade 1) | 33.3
  Hypertriglyceridemia (Grade 2) | 0
  Hypertriglyceridemia (Grade 3) | 33.3
  Hypertriglyceridemia (Grade 4) | 0
  Hyperuricemia (Grade 1) | 33.3
  Hyperuricemia (Grade 2) | 0
  Hyperuricemia (Grade 3) | 0
  Hyperuricemia (Grade 4) | 0

13. Secondary Outcome: Percentage of Participants Who Permanently Discontinued Idelalisib Due to a TEAE Beyond 28 Days of Idelalisib Exposure
Description: as for outcome 1
Time Frame: First dose date up to 30 days after last dose (up to approximately 3 years)
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Idelalisib
Number analyzed (Participants) | 6
percentage of participants | 16.7

ADVERSE EVENTS:
Time Frame: First dose date up to approximately 3 years
Description: The Full Analysis Set included all participants who took at least 1 dose of study drug.
Arm/Group | Idelalisib
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 5/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib (N=6)
Diarrhoea (Gastrointestinal disorders) | 3
Pyrexia (General disorders) | 1
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Transaminases increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib (N=6)
Anaemia (Blood and lymphatic system disorders) | 1
Optic disc haemorrhage (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Gastritis (Gastrointestinal disorders) | 3
Gastrointestinal pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Face oedema (General disorders) | 1
Fatigue (General disorders) | 1
Malaise (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 3
Vessel puncture site bruise (General disorders) | 1
Vessel puncture site inflammation (General disorders) | 1
Enteritis infectious (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 2
Infection (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Antithrombin III decreased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Transaminases increased (Investigations) | 2
Weight decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Renal failure (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years